CLINICAL TRIAL: NCT02143271
Title: A Single-dose Phase 1 Study of KHK7580 for Secondary Hyperparathyroidism in Patients Receiving Peritoneal Dialysis
Brief Title: Study of KHK7580 for Secondary Hyperparathyroidism in Patients Receiving Peritoneal Dialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7580-004
Record Dates: First submitted 2014-05-14; First posted 2014-05-21 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Secondary Hyperparathyroidism
Keywords: Secondary Hyperparathyroidism in Patients Receiving Peritoneal Dialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KHK7580 (Experimental)
  Interventions: Drug: KHK7580

INTERVENTIONS:
Drug: KHK7580 — Oral administration

SUMMARY:
This study is designed to evaluate safety, pharmacokinetics and pharmacodynamics after single administration of KHK7580 for secondary hyperparathyroidism in patients receiving peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Stable chronic renal disease patients receiving peritoneal dialysis for at least 16 weeks prior to the screening
* intact parathyroid hormone value ≥ 240 pg/mL at the screening
* Corrected serum calcium ≥ 8.4 mg/dL at the screening

Exclusion Criteria:

* Patients with primary hyperparathyroidism
* Patients who received cinacalcet within 2 weeks prior to the screening
* Patients who began to take or changed the dose/dosing regimen of active vitamin D/its analogs, phosphate binders and/or calcium containing compounds within 2 weeks prior to the screening
* Patients who underwent parathyroidectomy and/or parathyroid intervention
* Patients with uncontrolled hypertension and/or diabetes
* Patients with severe heart disorder
* Patients with severe hepatic disease
* Patients who take investigational drug in another clinical trial within 12 weeks prior to the screening
* Patients who have been judged ineligible to participate in the study by the investigator

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number and types of adverse events | For 8 days
  The safety of KHK7580 assessed by number and types of adverse events, laboratory tests, vital signs and electrocardiogram

SECONDARY OUTCOMES:
Profiles of pharmacokinetics | Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72 and 168 hours post-dose
  intact parathyroid hormone, whole parathyroid hormone, corrected serum calcium, phosphorus, intact fibroblast growth factor 23, ionized calcium, calcitonin

CONTACTS AND LOCATIONS:
Locations (1):
- Kyowa Hakko Kirin, Tokyo, Japan